CLINICAL TRIAL: NCT02255292
Title: A Study: Pure CBD as Single-agent for Solid Tumor.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Rotenberg Yakir, Hadas Lemberg, PhD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBD- HMO-CTIL
Record Dates: First submitted 2014-09-23; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cannabidiol (CBD) (Experimental): Patients with confirmed solid cancer, after progression of all the available standard therapy or unfit to standard therapy according to oncologist's view, measurable disease as determined by RECIST using CT, life expectancy of at least 6 months, Eastern Cooperative Oncology Group (ECOG) performance status < or = 2 and aged 18 years old and more will be included in the current study.
  Interventions: Drug: cannabidiol (CBD)

INTERVENTIONS:
Drug: cannabidiol (CBD) — Patients with confirmed solid cancer, after progression of all the available standard therapy or unfit to standard therapy according to oncologist's view, measurable disease as determined by RECIST using CT, life expectancy of at least 6 months, Eastern Cooperative Oncology Group (ECOG) performance status < or = 2 and aged 18 years old and more will be included in the current study

SUMMARY:
Increasing lines of evidence support an antitumourigenic effect of cannabinoids, including the cannabidiol (CBD) which does not posses the psychotropic effects of D9-tetrahydrocannabinol (THC). These include anti-proliferative and pro-apoptotic effects and they are known to interfere with several mechanisms in the tumorgenesis. Yet, evidence from clinical trials among cancer patients is needed. The aim of the current study is to evaluate the impact of CBD as single treatment among cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed solid cancer
* Approved license for using cannabis (from the ministry of health: Israel)
* Progression of all the available standard therapy / unfit to standard therapy according to oncologist's view
* Measurable disease as determined by RECIST
* Life expectancy of at least 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status < or = 2
* Aged 18 years old and more

Exclusion Criteria:

* Received cannabis therapy for any indication
* Previous systemic therapy of less than 3 weeks prior to and, if present, any acute toxicity > grade 1.
* Clinically significant cardiac disease or any history of psychosis
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate according to RECIST 1.1 | At baseline and at 8 weeks from time of first dose, by CT scans for RECIST 1.1
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response or partial response (CR+PR) as assessed by investigatorand RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Lemberg, PhD, Study Chair — Hadassah Medical Organization

REFERENCES:
- [Background] Mechoulam R, Peters M, Murillo-Rodriguez E, Hanus LO. Cannabidiol--recent advances. Chem Biodivers. 2007 Aug;4(8):1678-92. doi: 10.1002/cbdv.200790147. PMID 17712814